CLINICAL TRIAL: NCT04713358
Title: Effect of Nalmefene on the Quality of Resuscitation in Patients Under General Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Tong Ren Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-sx004
Record Dates: First submitted 2020-12-16; First posted 2021-01-19 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Resuscitation
Keywords: nalmefene; quality of resuscitation; general anesthesia
MeSH Terms: interventions — nalmefene; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nalmefene group (Experimental): for the nalmefene group, immediately Intravenous injection of Nalmefene (0.25 g/kg, plus normal saline to 1ml) after surgery
  Interventions: Drug: Nalmefene
- Control group (Placebo Comparator): Intravenous injection of normal saline 1ml immediately after surgery
  Interventions: Drug: normal Saline

INTERVENTIONS:
Drug: Nalmefene — Immediately Intravenous injection of Nalmefene (0.25 g/kg, plus normal saline to 1ml) after surgery
  Arms: Nalmefene group
Drug: normal Saline — Immediately Intravenous injection of normal saline 1ml after surgery
  Arms: Control group

SUMMARY:
Postoperative recovery is an important part of the patient's experience. A good recovery period is an important guarantee for the recovery of postoperative organs and functions after surgery. However, the delay in awakening after general anesthesia remains one of the biggest challenges facing anesthesiologists. The time of resuscitation depends on patient factors, effects of anesthetic factors, duration of surgery, and painful stimulation.

The delay of recovery after anesthesia was mainly caused by the use of anesthetic drugs during the perioperative period. The drugs commonly used during the perioperative period are opioid analgesics, sedatives and muscle relaxants. Studies have shown that intravenous opioids are more difficult to control than neuromuscular relaxants. Opioids can extend the recovery time after anesthesia by direct sedation of opioid receptors. It also reduces the sensitivity of brainstem chemoreceptors to carbon dioxide, leading to dose-dependent respiratory depression and hypercapnia, which affects the removal of volatile substances and carbon dioxide, and ultimately leads to coma. In addition, the active metabolites of some opioids can prolong the duration of action, especially in the case of impaired renal function, which can lead to delayed awakening.

As an opioid antagonist, nalmefene can inhibit or reverse the respiratory inhibition, sedation and hypotension effects of opioid drugs. Moreover, it has no opioid excitatory activity, does not produce respiratory inhibition, hallucinogenic effect or pupil dilation. In terms of inducing wakefulness during anesthesia, nalmefene can effectively reverse the sedative effect caused by opioids. There have been reports at home and abroad that nalmefene can be used to improve the effect of post-anesthesia resuscitation and reduce agitation during the waking period, but there is still a lack of large sample and well-designed randomized controlled studies to provide important data on how to improve the quality of anesthetized resuscitation. This study will conduct a rigorous randomized controlled studies,with large sample, and the research indicators for patients from the PACU roll-out to ordinary ward, using Aldrete score , in order to obtain a series of data of nalmefene used for anesthesia recovery , and to set the foundation of related research of nalmefene and similar drugs in clinical application in the future.

DETAILED DESCRIPTION:
Postoperative recovery is an important part of the patient's experience, regardless of the type of surgery. The recovery and prognosis of postoperative anesthesia have gradually become important indicators for judging the efficacy and quality of anesthesia. The recovery period of general anesthesia is an important transition period from anesthesia to wakefulness, and a good recovery period is an important guarantee for the recovery of postoperative organs and functions after surgery. However, the delay in awakening after general anesthesia remains one of the biggest challenges facing anesthesiologists. Postoperative resuscitation is the result of the removal of anesthetics from the brain. The time of resuscitation depends on patient factors, effects of anesthetic factors, duration of surgery, and painful stimulation.

The delay of recovery after anesthesia was mainly caused by the use of anesthetic drugs during the perioperative period. The drugs commonly used during the perioperative period are opioid analgesics, sedatives and muscle relaxants. Studies have shown that intravenous opioids are more difficult to control than neuromuscular relaxants. Opioids can extend the recovery time after anesthesia by direct sedation of opioid receptors. It also reduces the sensitivity of brainstem chemoreceptors to carbon dioxide, leading to dose-dependent respiratory depression and hypercapnia, which affects the removal of volatile substances and carbon dioxide, and ultimately leads to coma. In addition, the active metabolites of some opioids can prolong the duration of action, especially in the case of impaired renal function, which can lead to delayed awakening.

As an opioid antagonist, nalmefene can inhibit or reverse the respiratory inhibition, sedation and hypotension effects of opioid drugs. Moreover, it has no opioid excitatory activity, does not produce respiratory inhibition, hallucinogenic effect or pupil dilation. No pharmacological effects were observed without the administration of opioid agonists. In terms of inducing wakefulness during anesthesia, nalmefene can effectively reverse the sedative effect caused by opioids. There have been reports at home and abroad that nalmefene can be used to improve the effect of post-anesthesia resuscitation and reduce agitation during the waking period, but there is still a lack of large sample and well-designed randomized controlled studies to provide important data on how to improve the quality of anesthetized resuscitation. In order to speed up the awakening after anesthesia, promote the patients' consciousness and respiratory recovery, and improve the quality of awakening patients after anesthesia, the patients should control postoperative pain immediatly, improve the comfort of patients in the PACU, reduce the residence time of patients, speed up the circulation of operated patients, reduce the costs of PACU, and reduce the staff workload in the PACU. This study will conduct a rigorous randomized controlled studies, large sample, and the research indicators for patients from the PACU roll-out to ordinary ward, using Aldrete score , in order to obtain a series of data of nalmefene used for anesthesia recovery , and to lay the foundation of related research of nalmefene and similar drugs in clinical application in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Age is greater than or equal to 18 years old and less than 65 years old
2. Patients who need tracheal intubation under general anesthesia at the right time for orthopedics, urology, and thoracic elective surgery
3. Patients with American Society of Anesthesia physical status I or II
4. BMI≥18kg/m2, and ≤30kg/m2
5. The estimated anesthesia time is 1-4 hours.
6. The intraoperative narcotic analgesics (Sufentanil and Remifentanil)
7. The patient uses electronic intravenous analgesia pump after surgery
8. The patient has informed consent

Exclusion Criteria:

1. patients who refused to participate in the study
2. pantients who refuse intravenous analgesia
3. medical history or family history of cognitive disorders,delirium, epilepsy, abalienation, anxiety or depression;
4. recent use of anticholinergic drugs, antidepressants, antianxietics or anticonvulsants
5. medical history of organic brain diseases or cranial vascular diseases
6. patients with a history of allergy to any drug used in the study
7. History of drug addiction and alcoholic intemperance or drug abuse
8. The patient is diagnosed with severe heart and lung disease, or active heart disease, or severe hepatic dysfunction (ChildePugh class C), or severe renal dysfunction (undergoing dialysis before surgery) ,critical illness (preoperative ASA physical status classification > =3)
9. Participate in other clinical trials within 4 weeks
10. Patients who, during surgery, presented complications （cerebrovascular accidents、heart failure、pneumothorax）or transfer to the intensive care unit during hospitalization, and patients who chose to abandon.
11. Inability to communicate in the preoperative period because of coma, profound dementia, language barrier, or incapacity from severe disease
12. Anesthesia time is <1 hour or >4 hours
13. Patients had chronic pain (unsatisfied pain control for at least 1 month).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Time stay in PACU | From the end of the operation to the time that patient leave to inpatient ward up to 2hours
  The time between the end of the operation and the Aldrete score ≥9 in PACU

SECONDARY OUTCOMES:
Extube time | From the end of the operation to the time that patient leave to inpatient ward up to 2hours
  The time from the end of the operation to the removal of the endotracheal tube in PACU
Sedation - agitation score | From the end of the operation to the time that patient leave to inpatient ward up to 2hours
  Sedation - agitation score when the removal of the endotracheal tube
the directional force The time at which the Montreal score was ≥5 | From the end of the operation to the time that patient leave to inpatient ward up to 2hours
  The time at which the Montreal score was ≥5
Whether to use remedial analgesic drug (sufentanil) in PACU and the dosage | From the end of the operation to the time that patient leave to inpatient ward up to 2hours
  Whether to use remedial analgesic drug (fentanyl) in PACU and the dosage in PACU
VAS pain score (assessment time Aldrete score ≥9 points, 1h after surgery, 24h after surgery) | 1h after surgery, and 24h after surgery
  VAS pain score (assessment time Aldrete score ≥9 points, 1h after surgery, 24h after surgery) with assessment time Aldrete score ≥9 points, 1h after surgery, 24h after surgery)
The incidence of nausea and vomiting in PACU | From the end of the operation to the time that patient leave to inpatient ward up to 2hours
  The incidence of nausea and vomiting in PACU
Incidence of itch in PACU | From the end of the operation to the time that patient leave to inpatient ward up to 2hours
  Incidence of itch in PACU
Incidence of nausea and vomiting 0-24h after surgery | From the end of operation up to 24h after surgery
  Incidence of nausea and vomiting 0-24h after surgery
Incidence of pruritus 0-24h after surgery | From the end of operation up to 24h after surgery
  Incidence of pruritus 0-24h after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Weifeng Yu, Study Chair — Department of Anesthesiology, Renji Hospital, School of Medicine, SJTU
Locations (4):
- China (4):
  - The First Affiliated Hospital of Guangxi Medical University, Guangxi, Guangxi
  - Shanghai Tong Ren Hospital, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Zhengzhou University, Henan, Zhengzhou

REFERENCES:
- [Derived] Ma X, Liu J, Tang Y, Lian Q, Huai X, Liu W, Su D. The efficacy of nalmefene on anesthetic recovery of patients: a study protocol for a multicenter randomized controlled trial. Trials. 2023 Mar 1;24(1):156. doi: 10.1186/s13063-023-07169-4. PMID 36859316